CLINICAL TRIAL: NCT05507073
Title: A Comparison of Impingement Free Range of Motion With CT Scan After Manual and Robotic Total Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Royal Orthopaedic Hospital NHS Trust (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROH20ORTH16
Record Dates: First submitted 2022-06-27; First posted 2022-08-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Hip Osteoarthritis; Post-traumatic Osteoarthritis; Inflammatory Arthritis; Congenital Hip Problems; Avascular Necrosis of Hip
Keywords: hip replacement; THR; Robotic; Arthroplasty; Hip Surgery; Range of Motion
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: This will be a two-arm, single blind (assessor blind), randomised controlled group study. It will take place in the NHS hospital setting. Stratification will be performed for age and sex by means of a minimisation technique during randomisation for each subject entering the trial. Any participant that withdraws from the study will be replaced.
Who Masked: Outcomes Assessor
Masking Description: Individual/s carrying out assessment post-intervention are not aware of the intervention allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Total Hip Replacement (Active Comparator): Manual Total Hip Replacement
  Interventions: Procedure: Manual Total Hip Replacement
- Robot-Assisted Total Hip Replacement (Experimental): Robot-Assisted Total Hip Replacement
  Interventions: Procedure: Robot-Assisted Total Hip Replacement

INTERVENTIONS:
Procedure: Manual Total Hip Replacement — Implantation of a hip Device to alleviate pain and recover range of movement
  Other Names: Hip Arthroplasty; Hip Replacement; Total Hip Replacement
  Arms: Manual Total Hip Replacement
Procedure: Robot-Assisted Total Hip Replacement — Robot assisted Implantation of a hip Device to alleviate pain and recover range of movement
  Other Names: Hip replacement; Robotic Hip replacement; Robot Assisted Hip Arthroplasty
  Arms: Robot-Assisted Total Hip Replacement

SUMMARY:
Single-blinded randomised controlled trial comparing impingement with CT scan for manual and robotic total hip replacement. A pilot study of 50 participants.

DETAILED DESCRIPTION:
This will be a two-arm, single blind (assessor blind), randomised controlled group study. It will take place in the NHS hospital setting. Stratification will be performed for age and sex by means of a minimisation technique during randomisation for each subject entering the trial.

Arm 1: Manual total hip replacement with conventional templating Arm 2: Robotic total hip replacement In the study 25 participants will receive manual THR with conventional templating; the other 25 will receive Robotic THR.

Following recruitment in outpatient clinics, participants will undergo baseline assessments, including imaging and clinical assessment. All participants will then undergo THR surgery, which will likely entail an inpatient hospital stay of 1-2 days. Post-operative rehabilitation will be in line with the normal standard care for all participants. Post-operatively participants will make two visits to clinic at 6 weeks and 12 months (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or Female, aged 18 to 85 years at recruitment into trial
* Diagnosed with hip OA, post-traumatic OA, inflammatory arthropathy, , or congenital or developmental hip disease, avascular necrosis of the hip
* Listed for total hip replacement
* Suitable for Accolade 2 stem and Trident cup prostheses
* Female participants of child bearing potential must be willing to ensure that they use effective contraception during the trial
* In the Investigator's opinion, is able and willing to comply with all trial requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Inability to provide informed consent
* Previous surgery to the ipsilateral hip and implantation of metalwork.
* Significant co-morbidities that would make follow up difficult or uncomfortable
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Pregnancy or intention to become pregnant within the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Impingement analysis by a CT guided software in all participants to enable a comparison of post-operative impingement between robotic THR and manual THR | 6 weeks post-intervention
  To compare efficacy of Robotic THR in reducing post-operative impingement with Standard Manual THR

SECONDARY OUTCOMES:
Using the Forgotten Joint Score (FJS-12) to determine improvement in Patient reported outcome measures | 12 months
  To determine whether the Robotic THR improves patient reported outcome measures
Using the Oxford Hip score to determine improvement in Patient reported outcome measures | 12 months
  To determine whether the Robotic THR improves patient reported outcome measures
Using the EuroQol 5-D (EQ5-D) to determine improvement in Patient reported outcome measures | 12 months
  To determine whether the Robotic THR improves patient reported outcome measures
Measure leg length following surgery to determine whether robotic THR or manual THR is more effective at reducing leg length discrepancy. | 12 months
  To determine whether Robotic Surgery reduces leg length Discrepancy compared to manual THR
Measure the duration of surgery and compare the duration of robotic THR to manual THR | During Surgery
  To determine whether the Robotic THR increases operation duration compared to Manual surgery
Measure and compare the length of stay between Robotic and Manual THR surgeries | During length of stay in hospital average 3 days
  To determine if length of hospital stay is reduced after robotic THR .

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Orthopaedic Hospital NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No